CLINICAL TRIAL: NCT02933944
Title: A Non-Randomised Open-Label Phase Ib Exploratory Study of TG02-treatment as Monotherapy or in Combination With Pembrolizumab to Assess Safety and Immune Activation in Patients With Locally Advanced Primary and Recurrent Oncogenic RAS Exon 2 Mutant Colorectal Cancer
Brief Title: Exploratory Study of TG02-treatment as Monotherapy or in Combination With Pembrolizumab to Assess Safety and Immune Activation in Patients With Locally Advanced Primary and Recurrent Oncogenic RAS Exon 2 Mutant Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Changing priorities
Sponsor: Targovax ASA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT TG02-01
Record Dates: First submitted 2016-09-08; First posted 2016-10-14 (Estimated); Results first posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2019-06

CONDITIONS: Rectal Cancer
Keywords: locally recurrent
MeSH Terms: conditions — Rectal Neoplasms | interventions — pembrolizumab

ARMS (1):
- TG02-treatment (Experimental): Part I: The TG02-treatment consists of an intradermal injection of GM-CSF followed by an injection of TG02. The GM-CSF is to be given 15-30 minutes before TG02. TG02-treatment will be administered on Days 1, 8, 15, 22 and 36. If surgery after week 10, TG02-treatment will also be given at week 10 (Day 64).
  Part II: TG02-treatment will be given as described under Part I. In addition pembrolizumab will be administered.
  Interventions: Biological: TG02-treatment; Drug: Pembrolizumab

INTERVENTIONS:
Biological: TG02-treatment
Drug: Pembrolizumab

SUMMARY:
The purpose of this study is to determine safety and anti-tumor immune activation generated by TG02 and Granulocyte macrophage colony stimulating factor (GM-CSF), first as monotherapy (Part I), thereafter in combination with the checkpoint inhibitor pembrolizumab (Part II), in patients with locally advanced primary and recurrent colorectal cancer scheduled to have surgery.

Part I will include 4-6 patients and Part II will include up to 10 patients. Part I and Part II are separate and independent sequential components of the study. Patients will only be able to participate in either the Part I cohort or Part II cohort.

Main objective of the study is to investigate safety and immune response after TG02-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced primary and recurrent colorectal cancer (CRC) (histologically or cytologically confirmed adenocarcinoma), with a confirmed oncogenic KRAS exon 2, codon 12 or 13 mutations, eligible for radical pelvic surgery at time of enrolment.
* Patient is ≥18 years of age and able to consent
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Patient has adequate organ and bone marrow function within 28 days of study

  * Neutrophil count >1.5 x10^9/L
  * Platelets >100 x10^9/L
  * Hb >90g/L
  * Total bilirubin <1.5 upper limit of normal, ULN
  * ALT and AST <3.0 x ULN
  * Serum creatinine <3 x ULN or Creatinine Clearance ≥ 30ml/min (Cockroft-Gault or Nuclear GFR method)
  * PT and APTT <1.3 x ULN
* The patient is willing to provide study specific pre TG02-treatment biopsy of tumour mass and allow use of archival tumour biopsies. For patients where there are technical reasons a baseline biopsy cannot be performed but who fulfil all the other inclusion criteria, the investigator shall contact the medical monitor to discuss the possibility of including such patient.
* The patient is willing and able to comply with the protocol, and agrees to return to the hospital for study visits and examinations
* Men and women of childbearing potential must use adequate contraception to prevent pregnancy during the study. Adequate contraception is defined in the study as any medically recommended method (or combination of methods) as per standard of care. An adequate contraception includes hormonal contraception with implants or combined oral, transdermal or injectable contraceptives, certain intrauterine devices, bilateral tubal ligation, hysterectomy, or vasectomy of partner. A combination of male condom with either cap, diaphragm or sponge with spermicide are also considered acceptable. For women of childbearing potential a negative pregnancy test needs to be confirmed before inclusion.
* The patient has been fully informed about the study and is willing to participate in the study, and has provided written informed consent form prior to any trial specific screening procedures.

Exclusion Criteria:

* The patient has previously received an anticancer vaccine or immune checkpoint inhibitor, or participated in a trial involving the use of an anticancer vaccine or immune checkpoint inhibitor
* Patients where pre-surgery radiotherapy, chemotherapy or other anti-cancer therapy has not been completed ≥ 2 weeks prior to TG02-treatment
* The patients is receiving anti-cancer therapy for concurrent illness
* The patient has had a prior different malignancy within the last 3 years (excluding adequately treated basal cell or squamous cell carcinoma of the skin cancer, or localised low grade tumours considered cured and not requiring systemic therapy)
* The patient has uncontrolled or significant intercurrent or recent illness including:

  * auto-immune disorder or history of autoimmune disease requiring immunosuppressive treatment.
  * cardiac disorder such as uncontrolled cardiac failure, unstable angina or non-ST segment elevation myocardial infarction (NSTEMI) or myocardial infarction, uncontrolled arrhythmia less than 3 months before screening
  * stroke or thromboembolic event within 3 months of study commencement
  * active or uncontrolled severe infection
  * history of solid organ transplantation or any condition requiring chronic treatment with corticosteroids or other immunosuppressive agents
  * active coagulopathy/bleeding diathesis
  * cirrhosis, chronic active or untreated persistent hepatitis
  * history of adverse reactions to peptide vaccines
* The patient is pregnant or lactating.
* Has received an investigational drug within 4 weeks prior to study drug administration, or unless other has been agreed with the medical monitor
* Is currently receiving any agent with a known effect on the immune system, unless at dose levels that are not immunosuppressive (e.g. prednisone at 10 mg/day or less or as inhaled steroid at doses used for the treatment of asthma)
* Known history of positive tests for HIV/AIDS
* Are planned to receive yellow fever or other live (attenuated) vaccines during the course of study
* For Part II - any contraindication to receiving pembrolizumab:

If using the 50 mg lyophilized powder; hypersensitivity to the active substance (pembrolizumab) or to any of the excipients; L-histidine, L-histidine hydrochloride monohydrate, Sucrose, Polysorbate 80.

If using the 100 mg concentrate; hypersensitivity to the active substance (pembrolizumab) or to any of the excipients; L-histidine, Sucrose, Polysorbate 80

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-09; Primary Completion 2019-02 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (2):
  - Royal Brisbane & Women's Hospital (RBWH), Brisbane
  - Peter MacCallum Cancer Centre, Melbourne
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch

RESULTS

PARTICIPANT FLOW:
Groups:
- TG02-treatment: Part I: The TG02-treatment consists of an intradermal injection of GM-CSF followed by an injection of TG02. The GM-CSF is to be given 15-30 minutes before TG02. TG02-treatment will be administered on Days 1, 8, 15, 22 and 36. If surgery after week 10, TG02-treatment will also be given at week 10 (Day 64).
  Part II: TG02-treatment will be given as described under Part I. In addition pembrolizumab will be administered. Part II was not conducted.
Period: Overall Study
Arm/Group | TG02-treatment
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TG02-treatment
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 1
  Australia | 5

OUTCOME MEASURES:

1. Primary Outcome: Patients Safety During Study
Description: Safety of TG02-treatment by assessment of laboratory parameters (routine haematology and biochemistry), vital signs and recording of adverse events
Time Frame: From start of study until End of study, which is approximately 4 weeks after surgery and maximum 20 weeks after start of TG02-treatment
Measure: Number; unit: Participants
Groups:
- TG02-treatment: Part I: The TG02-treatment consists of an intradermal injection of GM-CSF followed by an injection of TG02. The GM-CSF is to be given 15-30 minutes before TG02. TG02-treatment will be administered on Days 1, 8, 15, 22 and 36. If surgery after week 10, TG02-treatment will also be given at week 10 (Day 64).
  Part II: TG02-treatment will be given as described under Part I. In addition pembrolizumab will be administered.
  TG02-treatment
  Pembrolizumab
Arm/Group | TG02-treatment
Number analyzed (Participants) | 6
Participants
  Number of patients with Treatment Emergent Adverse Events (TEAEs) | 6
  Number of patients with Treatment Emergent Adverse Serious Event (TESAE) | 2
  Number of patients with Grade 3 or 4 Treatment Emergent Adverse Event (TEAE) | 2
  Number of patients with Treatment Emergent Adverse Event related to any of the study treatments | 3
  Number of patients with fatal events | 0
  Number of patients discontinuing for Adverse Events | 0

2. Primary Outcome: Patients' Immune Response Assessed by Delayed Type Hypersensitive (DTH) Test
Description: Number of patients with systemic TG02 specific immune response assessed by a Delayed Type Hypersensitivity (DTH) test
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | TG02-treatment
Number analyzed (Participants) | 6
Participants | 4

3. Primary Outcome: Systemic Immune Response: T-cell Response
Description: Systemic immune response assessed as change in presence of TG02 specific T-cells in peripheral blood
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | TG02-treatment
Number analyzed (Participants) | 6
Participants | 3

4. Primary Outcome: Immunological Activation in Tumour Mass by Assessing Number of Patients With Increased Intra-tumoural Lymphocytes.
Description: Immunological activation in tumour mass by assessing fold changes from baseline of intra-tumoural lymphocytes.
Time Frame: 8 weeks
Population: Due to insufficient number of baseline samples, no valid results can be derived i.e. change in number of activated intratumoural lymphocytes from baseline.
Groups:
- TG02-treatment: Part I: The TG02-treatment consists of an intradermal injection of GM-CSF followed by an injection of TG02. The GM-CSF is to be given 15-30 minutes before TG02. TG02-treatment will be administered on Days 1, 8, 15, 22 and 36. If surgery after week 10, TG02-treatment will also be given at week 10 (Day 64).
Arm/Group | TG02-treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Change of Immune Suppression Factors e.g. PD-1 and T-reg From Pre to Post Treatment
Description: Number of patients with changes from baseline in immune suppression factors (such as PDL1, Treg and MSDC) from tumour samples collected pre TG02/GMCSF treatment
Time Frame: 8 weeks
Population: Due to the low number of baseline samples, no treatment effect can be concluded.
Arm/Group | TG02-treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in Pathological Responses and Markers of Apoptosis in Tumour Tissue
Time Frame: 8 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Changes in Standard Uptake Values (SUV) Will be Assessed by FDG PET-CT Images
Time Frame: From screening until surgery
Reporting Status: Not Posted

8. Secondary Outcome: Changes in the Tumour Marker Carcinoembryonic Antigen (CEA) Throughout Treatment Will be Assessed by Analysis of Blood Samples to Follow the Evolution of Disease Under Treatment
Time Frame: From screening until surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 14 to 20 weeks on study with up to 10 weeks of treatment
Arm/Group | TG02-treatment
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TG02-treatment (N=6)
Urinary tract infection (Infections and infestations) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TG02-treatment (N=6)
Influenza like illness (General disorders) | 2 (4)
Chills (General disorders) | 1 (4)
Injection site pain (General disorders) | 1 (1)
Injection site pruritus (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (2)
Pyrexia (General disorders) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (2)
Laryngitis (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT02933944/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT02933944/SAP_001.pdf